CLINICAL TRIAL: NCT05384522
Title: Analysis of the Prognostic Role of Epigenetic Biomarkers in Relation to the Motor Decline in Parkinson's Disease
Acronym: BioGenPark
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Other Study IDs: INRCA_002_2022
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; aging; biomarkers; DNA methylation; precision medicine; epigenomics; genetics; disease progression
MeSH Terms: conditions — Parkinson Disease; Disease Progression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A volume of approximately 35 mL (5ml EDTA tubes, 5ml LiHep tubes, 10 ml serum tubes, 10 ml whole blood tubes and 5 ml citrate tubes) of peripheral blood will be collected at baseline and after 6 and 12 months. The buffy coat for DNA extraction will be stored from the same tubes. Five mL of urine will be collected from all study participants at baseline and at 6 and 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's Disease subjects: Subjects with Parkinson Disease aged 65 years or more at Hoehn and Yahr stage ≤3
  Interventions: Other: blood samples collection

INTERVENTIONS:
Other: blood samples collection — Blood samples will be drawn at baseline and at 6 and 12 months from baseline

SUMMARY:
BioGenParkinson is an observational, prospective cohort study evaluating biomarkers of Parkinson's Disease (PD) progression in community-dwelling subjects aged 65 years or more, consecutively referring to INRCA outpatient clinic of the Neurology Unit. Selected patients will undergo clinical and laboratory evaluations at the baseline, and will be followed up after 6 and 12 months. The biological evaluation will include the determination of i) routine biological parameters ii) advanced biomarkers such as epigenetic analysis of DNA methylation, genetic analysis on multiple loci associated with PD progression and specific proteins associated with motor and non-motor decline. After obtaining all data, multiple statistical analysis will be performed to evaluate the most accurate prognostic biomarkers of PD progression at this stage of disease.

DETAILED DESCRIPTION:
The objective of the BioGenParkinson study is the evaluation of the prognostic accuracy of epigenetic, genetic and protein biomarkers in relation to Parkinson's Disease (PD) motor symptoms progression (assessed by changes in Unified Parkinson's Disease Rating Scale Part III (UPDRS III)) in biological samples of 103 PD patients aged 65 or more. Changes of quality of life (assessed by Parkinson's Disease Questionnaire 39 item (PDQ-39)) and cognitive performance (assessed by the Mini-Mental State Examination (MMSE)) will be also investigated. The characterization of the PD patients' phenotypes and genotypes will allow the investigation on the predisposition to a severe progression of the disease, in order to early predict the progression of the disease and improving the accuracy of personalized interventions. The evidence collected will inform multidisciplinary and personalized interventions in the future.

Among the advanced biomarkers that will be evaluated in the Study, epigenetic analysis of CpG loci such as cg17445913 in KCNB1 gene, cg02920897 in DLEU2 gene and cg01754178 in PTPRN2 gene are expected to improve the prognostic accuracy of motor and cognitive decline of PD patients at Hoehn and Yahr stage II/III after 12 months of follow up. Genetic analysis in purified genomic DNA samples will be performed on multiple loci associated with PD progression such as rs2230288 and rs75548401 in order to confirm their association with motor decline over time, and to assess their association with non-motor decline.

Protein analysis on bone sialoprotein (BSP), osteomodulin (OMD), aminoacylase-1 (ACY1), and growth hormone receptor (GHR) will be also evaluated with respect to motor and non-motor decline in PD patients in order to be compared with the other biomarkers. Scores on UPDRS Parts III, obtained by using using the published cut-offs classification of MDS-UPDRS severity, will be drawn at the baseline, at 6-month and at 12-month follow-up visits, in order to assess PD motor progression. Additional assessments include demographic and clinical data, Parkinson Disease Questionnaire 39 item (PDQ-39) Hoehn and Yahr stage, MMSE, Frontal Assessment Battery (FAB), list of disease and medication, falls, functional status, quality of life and socio-economic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* PD at Hoehn and Yahr stage ≤3
* MMSE test ≥24 score

Exclusion Criteria:

* MMSE score < 24
* Severe cardiovascular diseases (including congestive heart failure NYHA=4, acute coronary syndrome, stroke)
* History of traumatic brain injury, previous deep brain surgery
* Current substance or alcohol abuse
* Reduced life expectancy less than six months

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Community-dwelling subjects aged 65 years or more with Parkinson Disease at Hoehn and Yahr stage ≤3
Sampling Method: Non-Probability Sample
Enrollment: 103 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Prognostic role of epigenetic biomarkers with respect to the advancing of PD motor decline | Baseline and 12 months later
  Change of Unified Parkinson's Disease Rating Scale (UPDRSIII) in relation to the baseline methylation status of the following epigenetic biomarkers: CpG loci cg17445913, cg02920897 and cg01754178. PD motor decline will be defined by an increase of UPDRS III at least of 2.4 points/year.

SECONDARY OUTCOMES:
Prognostic role of genetic biomarkers with respect to the advancing of PD motor decline | Baseline and 12 months later
  Change of Unified Parkinson's Disease Rating Scale (UPDRSIII) in relation to the presence of mutations of the GBA coding variants rs2230288 and rs75548401. PD motor decline will be defined by an increase of UPDRS III at least of 2.4 points/year.
Prognostic role of bone sialoprotein (BSP) with respect to the advancing of PD motor decline | Baseline and 12 months later
  Change of Unified Parkinson's Disease Rating Scale (UPDRSIII) in relation to the levels of baseline bone sialoprotein (BSP). PD motor decline will be defined by an increase of UPDRS III at least of 2.4 points/year.
Prognostic role of osteomodulin (OMD) with respect to the advancing of PD motor decline | Baseline and 12 months later
  Change of Unified Parkinson's Disease Rating Scale (UPDRSIII) in relation to the levels of baseline osteomodulin (OMD).
Prognostic role of aminoacylase-1 (ACY1) with respect to the advancing of PD motor decline | Baseline and 12 months later
  Change of Unified Parkinson's Disease Rating Scale (UPDRSIII) in relation to the levels of baseline aminoacylase-1 (ACY1).PD motor decline will be defined by an increase of UPDRS III at least of 2.4 points/year.
Prognostic role of growth hormone receptor (GHR) with respect to the advancing of PD motor decline | Baseline and 12 months later
  Change of Unified Parkinson's Disease Rating Scale (UPDRSIII) in relation to the levels of baseline growth hormone receptor (GHR).PD motor decline will be defined by an increase of UPDRS III at least of 2.4 points/year.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pelliccioni, MD, Principal Investigator — IRCCS INRCA, Ancona, Italy